CLINICAL TRIAL: NCT06426693
Title: Connectome-based Neurofeedback of the Craving Network to Reduce Food Cue Reactivity
Brief Title: Craving Network Neurofeedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000037084; 1R01DK136623-01A1 (NIH)
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback (Experimental): Three imaging (fMRI) sessions of experimental feedback.
  Interventions: Device: Experimental feedback
- Control neurofeedback (Sham Comparator): Three imaging (fMRI) sessions of sham feedback.
  Interventions: Device: Control feedback

INTERVENTIONS:
Device: Experimental feedback — Participants provided with feedback of target brain activation patterns (e.g., thermometer) and will be instructed to try to change the feedback (e.g., decrease the thermometer).
  Arms: Neurofeedback
Device: Control feedback — Participants provided with control (sham, yoked to another participant) feedback (e.g., thermometer) and will be instructed to try to change the feedback (e.g., decrease the thermometer).
  Arms: Control neurofeedback

SUMMARY:
This project tests whether individuals with overweight or obesity and high craving can learn to change their brain response to food cues using neurofeedback, to impact their craving and eating behavior.

DETAILED DESCRIPTION:
Aim 1 of this study is to test whether neurofeedback from the craving network is associated with reduced craving network strength.

Aim 2 of this study is to test whether neurofeedback from the craving network is associated with reduced food craving and changes in eating behavior.

Aim 3 of this study is to test whether neurofeedback from the craving network is associated with changes in resting state functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 60 years
* Body mass index >25 kg/m2
* >2.37 Food Craving Inventory score

Exclusion Criteria:

* Current or past 6 months use of anti-obesity medications
* Weight-reduced state defined as >10% weight reduction in the past 6 months.
* Nicotine use
* Current diagnosis of neurological or psychiatric disorder
* Obesity-related diseases such as type-2 diabetes
* Contraindications to MRI
* Baseline scanning with motion >0.15mm frame to frame displacement.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in craving network strength during transfer runs | Week 1 and 3
  Craving network strength will be measured during transfer (i.e., no feedback) runs and compared across scan sessions.
Change in Food Craving Inventory Mean Score | Week 1, Week 7
  Food Craving Inventory has 28 items rated 1-5 and overall mean is calculated, range 1-5 with higher score indicating higher craving. FCI will be compared between baseline and 1 month follow-up.
Change in Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool Healthy Eating Index (HEI). | Week 1, Week 7
  ASA-24 HEI is scored 0-100 with 100 indicating healthier diet and composite scores examined to interpret the overall score. HEI will be compared between baseline and 1 month follow-up.
Change in craving network strength during resting state runs | Week 1 and 3
  Craving network strength will be measured during resting state runs and compared across scan sessions.
Change in Food Rating Task healthiness, tastiness, and choice scores | Week 1, Week 7
  Food Rating Task outcomes include healthiness, tastiness, and choice. Healthiness and tastiness mean score is taken, range 1-5, with 5 indicating higher healthiness or tastiness. Choice is counted from 0-48 items choosing the food item over the neutral reference food item, with higher values indicating more frequent choice. Food Ratings will be compared between baseline and 1 month follow-up.
Change in Food Snack Task caloric intake | Week 1 and 3
  Food Snack Task will be used to measure caloric intake (out of a maximum value to calories offered) and compared across scan sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Garrison, PhD, Principal Investigator — Yale University
Locations (1):
- Yale MRRC Anlyan Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be findable for the research community through OpenNeuro and NITRC search functions.
Time Frame: The research community will have access to data when the award ends.